CLINICAL TRIAL: NCT07212387
Title: Effectiveness of Sacral Neuromodulation in Patients With Coexisting Faecal and Urinary Incontinence ("Double Incontinence")
Brief Title: Sacral Neuromodulation in Patients With Double Incontinence
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FNO-Urology-DI
Record Dates: First submitted 2025-09-30; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Double Incontinence; Faecal Incontinence; Urinary Incontinence
Keywords: Double incontinence; Faecal incontinence; Urinary incontinence; Sacral neurostimulation
MeSH Terms: conditions — Encopresis; Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: The study subjects will be enrolled in one experimental group
Masking Description: No masking is being used in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sacral neuromodulation (Experimental): Female patients with double incontinence (DI) will be enrolled into this study group. The study subjects will undergo sacral neurostimulation (SNM).
  Interventions: Procedure: Sacral neurostimulation

INTERVENTIONS:
Procedure: Sacral neurostimulation — Sacral neurostimulation (SNS), or sacral neuromodulation (SNM), is a minimally invasive, reversible treatment for bladder and bowel control problems, including overactive bladder and fecal incontinence.

SUMMARY:
This is a prospective study evaluating the effect of a treatment method of sacral neuromodulation (SNM), the use of which is approved and recommended for the treatment of both faecal incontinence (FI) and urinary incontinence (UI). A new aspect of the study is monitoring the effect of SNM in patients with both types of incontinence (faecal and urinary) occurring simultaneously. The study will use diagnostic methods and procedures that are part of the usual examination algorithm. The study will not impose any burden on patients beyond the scope of routine examination and treatment procedures.

DETAILED DESCRIPTION:
Faecal incontinence (FI) is defined as the involuntary loss of solid or liquid stool in patients. Incontinence harms the patient psychologically, socially and medically. FI is associated with an increased incidence of various skin conditions and inflammatory diseases, including multiple urinary tract infections.

Treatment of FI usually begins with non-invasive strategies such as dietary and lifestyle changes, physiotherapy with biofeedback, and pharmacotherapy. If conservative methods do not improve symptoms, surgical options are considered, such as sphincter reconstruction, anal sphincter augmentation, and artificial sphincter. Neurostimulation methods, including sacral neuromodulation (SNM), are another option.

Participation in the study will be offered to patients with proven DI who have failed primary conservative treatment. Eligible patients will be indicated to perform the 1st phase of SNM, which consists of inserting a stimulating electrode into the sacral root area and connecting it to an external stimulation source according to the standard procedure [21].

After 2 weeks of stimulation in the test phase, its effectiveness will be evaluated. A positive treatment response is defined as:

An improvement of more than 50% in any of the DI symptoms (according to the bladder and bowel diary in 3 days or 7 days, respectively) and the patient also rates the improvement of her condition as 1 ("very much improved") or 2 ("much improved") using the PGI-I scale An improvement of at least 2 DI symptoms by more than 25% (according to the bladder and bowel diary in 3 days or 7 days, respectively) and the patient also rates the improvement of her condition as 1 ("very much improved") or 2 ("much improved") using the PGI-I scale If the patient achieves a positive treatment response at the end of the test phase, she will be indicated for the 2nd phase of SNM, during which the external stimulation source will be replaced by an implanted stimulation generator. The patient will then continue to be monitored 3, 6 and 12 months after implantation. This will terminate the patient's participation in the study and they will continue to receive treatment or follow-up according to the current clinical recommendations for the treatment of FI and UI.

If the patient does not achieve a positive treatment response at the end of the test phase, the electrode and external stimulator will be removed, the patient will be excluded from the study and will be further monitored or treated according to the current clinical recommendations for the treatment of FI and UI.

Urinary incontinence (UI) is defined as any involuntary leakage of urine. UI has a major impact on the quality of life of affected patients, as well as clearly documented health and socioeconomic consequences.

Conservative (pelvic floor muscle training), semi-invasive (application of so-called "bulking agents" into the urethra) and surgical methods (implantation of tension-free homologous or heterologous bands under the urethra) are used in the treatment of female stress incontinence.

Pharmacotherapy is mainly used in the treatment of urge incontinence. In those patients in whom it is not sufficiently effective or is accompanied by adverse effects, treatment with botulinum toxin applied to the bladder wall or various neuromodulation methods is recommended.

Coexistent fecal and urinary incontinence (double incontinence - DI) is a condition in which symptoms of FI and UI are expressed simultaneously.

Given its high prevalence, DI represents a significant cost to society and healthcare systems. Patients with DI face a number of significant problems that affect their physical (skin irritation and infection, unpleasant odour, hygiene problems, insufficient sleep, etc.) and psychological health (anxiety and depression, social isolation, disrupted relationships, etc.) and quality of life.

Therefore, the treatment of DI is very complex, multidisciplinary and it is very difficult to create uniform clinical recommendations.

Sacral nerve stimulation (SNS) delivers painless electrical impulses to the sacral nerves to improve pelvic organ function. Currently approved indications include urge urinary incontinence, non-obstructive urinary retention, and faecal incontinence. Further studies investigating the treatment outcomes of SNS in patients with DI are therefore highly desirable and needed.

Investigational tools used during the study Patient global impression of improvement (PGI-I) - is a simple screening tool that was created to assess the effect of treatment on a given pathological condition. It is a Likert scale with a rating from 1 ("very much improvement") to 7 ("very much deterioration").

Bladder and bowel diary - is a basic screening tool for assessing the severity of urinary and faecal incontinence symptoms. The patient records data on the time and amount of fluids consumed and data on the time and volume of urine excreted in the diary. She also adds data on the number of episodes of urgency and urinary incontinence. Similarly, she records the number of defecations and data on the number of episodes of urgency and faecal incontinence. The patient records data on urination for 3 days, data on stool for a total of 7 days.

The Wexner Questionnaire - Wexner Score, is a widely used and recognized tool for assessing the severity of faecal incontinence. It serves to objectify and quantify symptoms, which is crucial for diagnosing, monitoring progression, and evaluating the effectiveness of FI treatment. The Wexner Score focuses on five key parameters related to faecal incontinence: gas leakage, liquid stool leakage, solid stool leakage, wearing pads/protective devices, and lifestyle changes. Each of these five parameters is scored on a scale from 0 to 4, where 4 is the worst, and the maximum possible score is 20 points - indicating complete faecal incontinence.

The Faecal Incontinence Quality of Life Scale (FIQL) is a specific quality of life questionnaire designed to assess the impact of FI on various aspects of a patient's life. Unlike incontinence severity scores (such as the Wexner or St. Mark's scores), which only quantify the frequency and type of leakage, the FIQL focuses on how incontinence affects the patient's daily life, psychological well-being, and social interactions. Patients typically rate their feelings or the frequency of the problems on a Likert scale (from 1 to 5, with higher numbers indicating better quality of life or less impact).

The International Consultation of Incontinence Questionnaire - Urinary Incontinence short form (ICIQ-UI SF) is one of the most commonly used tools to assess the effectiveness of interventions in functional urology. This validated questionnaire consists of 3 questions that assess the frequency, severity, and overall impact of incontinence on quality of life. The total score can range from 0-21, with higher scores indicating greater severity of urinary incontinence.

The International Consultation of Incontinence-Overactive Bladder (ICIQ-OAB) is a validated questionnaire used to assess the effectiveness of treatment for urge incontinence and overactive bladder. It consists of 4 questions, focusing on the main symptoms of frequency, nocturia, urgency and urge incontinence. Each question has a sub-question assessing the impact of a specific symptom on quality of life. The total symptom score can be 0-16, the impact score on quality of life can take values of 0-40. In both cases, the higher the score, the greater the severity of urinary incontinence and the greater the negative impact on quality of life.

The Incontinence - Quality of Life (I-QoL) questionnaire is a validated questionnaire assessing the impact of urinary incontinence on patients' quality of life. It consists of 22 questions that the patient answers using a Likert scale from 1 ("Always") to 5 ("Never"). The higher the total score, the better the quality of life, or the smaller the impact of incontinence on quality of life.

Monitoring of the number and severity of treatment-related adverse events (TRAE) will be carried out according to Good Clinical Practice standards.

ELIGIBILITY:
Inclusion Criteria:

* Adult women over 18 years of age
* Consent to participate in the study
* Willingness to undergo examination, treatment and follow-up according to the protocol
* DI symptoms characterized by:
* Grade III fecal incontinence (patient is unable to consciously hold in wind, loose or hard stools)
* At least 2 episodes of fecal incontinence during the week (according to bladder and bowel diary)
* At least 1 episode of involuntary urine leakage per day (according to bladder and bowel diary)
* Total score of the ICIQ-UI SF questionnaire
* DI symptoms for more than 6 months
* Failure of previous conservative treatment

Exclusion Criteria:

* Rapidly progressing neurological diseases
* Known severe congenital malformations of the anorectum and/or lower urinary tract
* Presence of a foreign body in the urinary tract - urolithiasis, urinary catheter, ureteral stent
* Pregnancy, lactation
* Active urinary tract infection
* Active malignant disease
* Clinically significant pelvic organ prolapse
* Active inflammatory bowel disease (Crohn's disease, ulcerative colitis)
* In the case of an associated lesion of the external anal sphincter, a defect greater than 90 degrees
* Previous pelvic radiotherapy less than 12 months prior to study enrolment
* Previous pelvic organ descent surgery less than 12 months prior to study enrolment
* Previous stress urinary incontinence surgery less than 12 months prior to study enrolment
* Previous childbirth less than 12 months prior to study enrollment
* Anatomical malformations of the sacrum that preclude implantation of the SNM electrode
* Low patient compliance
* Inability to control the neurostimulator

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study is intended for female patients with double incontinence only.
Enrollment: 30 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2029-11 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Overall effect of SNM | 18 months
  Evaluation of the overall effect of SNM in patients with DI from the patient's perspective using the so-called "patients reported outcome measures" (PROM) with the Patient Global Impression - Improvement questionnaire will be performed.

SECONDARY OUTCOMES:
The number of responders at the end of the test phase | 2 weeks for the patient, 4 years for the investigator
  The number of responders at the end of the test phase will be observed
Bladder and bowel diary - the number of FI episodes | 3 and 7 days
  The number of FI episodes from the bladder and bowel diary will be observed for the monitored period of 3 and 7 days
Bladder and bowel diary - the number of faecal urgency episodes | 3 and 7 days
  The number of faecal urgency episodes from the bladder and bowel diary will be observed for the monitored period of 3 and 7 days
Bladder and bowel diary - the number of UI episodes | 3 and 7 days
  The number of UI episodes from the bladder and bowel diary will be observed for the monitored period of 3 and 7 days
Bladder and bowel diary - the number of urinary urgency episodes | 3 and 7 days
  The number of urinary urgency episodes from the bladder and bowel diary will be observed for the monitored period of 3 and 7 days
Wexner questionnaire total score | 18 months for the patient, 4 years for the investigator
  The Wexner questionnaire total score will be observed and recorded
FIQL questionnaire total score | 18 months for the patient, 4 years for the investigator
  The FIQL (Faecal Incontinence Quality of Life Scale) questionnaire total score will be observed and recorded
ICIQ-SF questionnaire total score | 18 months for the patient, 4 years for the investigator
  The ICIQ-SF (International Consultation of Incontinence Questionnaire) questionnaire total score will be observed and recorded
ICIQ-OAB questionnaire total score | 18 months for the patient, 4 years for the investigator
  The ICIQ-OAB (International Consultation on Incontinence Questionnaire - Overactive Bladder) questionnaire total score will be observed and recorded
I-QoL questionnaire total score | 18 months for the patient, 4 years for the investigator
  The I-QoL (Incontinence - Quality of Life ) questionnaire total score will be observed and recorded
Number and severity of treatment-related adverse events (TRAE) | 18 months for the patient, 4 years for the investigator
  The number and severity of treatment-related adverse events (TRAE) will be observed and recorded

CONTACTS AND LOCATIONS:
Overall Officials: Milan Tesař, MD, Ph.D., Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No
There is no plan to make the individual participant data available to other researchers. The data may be provided upon reasonable request.

REFERENCES:
- [Background] Wagner TH, Patrick DL, Bavendam TG, Martin ML, Buesching DP. Quality of life of persons with urinary incontinence: development of a new measure. Urology. 1996 Jan;47(1):67-71; discussion 71-2. doi: 10.1016/s0090-4295(99)80384-7. PMID 8560665
- [Background] Jackson S, Donovan J, Brookes S, Eckford S, Swithinbank L, Abrams P. The Bristol Female Lower Urinary Tract Symptoms questionnaire: development and psychometric testing. Br J Urol. 1996 Jun;77(6):805-12. doi: 10.1046/j.1464-410x.1996.00186.x. PMID 8705212
- [Background] Lim R, Liong ML, Lim KK, Leong WS, Yuen KH. The Minimum Clinically Important Difference of the International Consultation on Incontinence Questionnaires (ICIQ-UI SF and ICIQ-LUTSqol). Urology. 2019 Nov;133:91-95. doi: 10.1016/j.urology.2019.08.004. Epub 2019 Aug 12. PMID 31415780
- [Background] Jorge JM, Wexner SD. Etiology and management of fecal incontinence. Dis Colon Rectum. 1993 Jan;36(1):77-97. doi: 10.1007/BF02050307. PMID 8416784
- [Background] Sultan AH, Monga A, Lee J, Emmanuel A, Norton C, Santoro G, Hull T, Berghmans B, Brody S, Haylen BT. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female anorectal dysfunction. Neurourol Urodyn. 2017 Jan;36(1):10-34. doi: 10.1002/nau.23055. Epub 2016 Oct 22. PMID 27770550
- [Background] Matzel KE, Chartier-Kastler E, Knowles CH, Lehur PA, Munoz-Duyos A, Ratto C, Rydningen MB, Sorensen M, van Kerrebroeck P, de Wachter S. Sacral Neuromodulation: Standardized Electrode Placement Technique. Neuromodulation. 2017 Dec;20(8):816-824. doi: 10.1111/ner.12695. Epub 2017 Oct 4. PMID 28975677
- [Background] Chodez M, Trilling B, Thuillier C, Boillot B, Barbois S, Faucheron JL. Results of sacral nerve neuromodulation for double incontinence in adults. Tech Coloproctol. 2014 Dec;18(12):1147-51. doi: 10.1007/s10151-014-1231-z. Epub 2014 Nov 8. PMID 25380739
- [Background] Duelund-Jakobsen J, Lehur PA, Lundby L, Wyart V, Laurberg S, Buntzen S. Sacral nerve stimulation for faecal incontinence - efficacy confirmed from a two-centre prospectively maintained database. Int J Colorectal Dis. 2016 Feb;31(2):421-8. doi: 10.1007/s00384-015-2411-7. Epub 2015 Oct 21. PMID 26490052
- [Background] Wexner SD, Coller JA, Devroede G, Hull T, McCallum R, Chan M, Ayscue JM, Shobeiri AS, Margolin D, England M, Kaufman H, Snape WJ, Mutlu E, Chua H, Pettit P, Nagle D, Madoff RD, Lerew DR, Mellgren A. Sacral nerve stimulation for fecal incontinence: results of a 120-patient prospective multicenter study. Ann Surg. 2010 Mar;251(3):441-9. doi: 10.1097/SLA.0b013e3181cf8ed0. PMID 20160636
- [Background] Kaiser AM, Orangio GR, Zutshi M, Alva S, Hull TL, Marcello PW, Margolin DA, Rafferty JF, Buie WD, Wexner SD. Current status: new technologies for the treatment of patients with fecal incontinence. Surg Endosc. 2014 Aug;28(8):2277-301. doi: 10.1007/s00464-014-3464-3. Epub 2014 Mar 8. PMID 24609699
- [Background] Brazzelli M, Murray A, Fraser C. Efficacy and safety of sacral nerve stimulation for urinary urge incontinence: a systematic review. J Urol. 2006 Mar;175(3 Pt 1):835-41. doi: 10.1016/S0022-5347(05)00326-5. PMID 16469561
- [Background] Noblett KL, Cadish LA. Sacral nerve stimulation for the treatment of refractory voiding and bowel dysfunction. Am J Obstet Gynecol. 2014 Feb;210(2):99-106. doi: 10.1016/j.ajog.2013.07.025. Epub 2013 Jul 27. PMID 23899452
- [Background] Baudouin C, Simitzis-Le Flohic AM, Peirone D, Le Fichoux Y, Gastaud P. [Acanthamoeba keratitis in subjects with contact lenses]. Presse Med. 1990 Nov 17;19(38):1759-61. French. PMID 2147501
- [Background] Meschia M, Buonaguidi A, Pifarotti P, Somigliana E, Spennacchio M, Amicarelli F. Prevalence of anal incontinence in women with symptoms of urinary incontinence and genital prolapse. Obstet Gynecol. 2002 Oct;100(4):719-23. doi: 10.1016/s0029-7844(02)02215-9. PMID 12383540
- [Background] Gonzalez-Argente FX, Jain A, Nogueras JJ, Davila GW, Weiss EG, Wexner SD. Prevalence and severity of urinary incontinence and pelvic genital prolapse in females with anal incontinence or rectal prolapse. Dis Colon Rectum. 2001 Jul;44(7):920-6. doi: 10.1007/BF02235476. PMID 11496068
- [Background] Cameron AP, Chung DE, Dielubanza EJ, Enemchukwu E, Ginsberg DA, Helfand BT, Linder BJ, Reynolds WS, Rovner ES, Souter L, Suskind AM, Takacs E, Welk B, Smith AL. The AUA/SUFU guideline on the diagnosis and treatment of idiopathic overactive bladder. Neurourol Urodyn. 2024 Nov;43(8):1742-1752. doi: 10.1002/nau.25532. Epub 2024 Jul 15. PMID 39010271
- [Background] Ruffolo AF, Frigerio M, Barba M, Salvatore S, Athanasiou S, Espuna-Pons M, Serati M. European Urogynaecological Association Position Statement: Implantable Devices for Female Stress Incontinence Surgery. Eur J Obstet Gynecol Reprod Biol. 2025 May;309:175-185. doi: 10.1016/j.ejogrb.2025.03.049. Epub 2025 Mar 25. PMID 40157225
- [Background] Luo C, Niu X. A comprehensive review of conservative therapies for female stress urinary incontinence: Advancements, efficacy, and future directions. Curr Urol. 2025 Mar;19(2):84-89. doi: 10.1097/CU9.0000000000000270. Epub 2025 Jan 21. PMID 40314017
- [Background] Lukacz ES, Santiago-Lastra Y, Albo ME, Brubaker L. Urinary Incontinence in Women: A Review. JAMA. 2017 Oct 24;318(16):1592-1604. doi: 10.1001/jama.2017.12137. PMID 29067433
- [Background] Patel UJ, Godecker AL, Giles DL, Brown HW. Updated Prevalence of Urinary Incontinence in Women: 2015-2018 National Population-Based Survey Data. Female Pelvic Med Reconstr Surg. 2022 Apr 1;28(4):181-187. doi: 10.1097/SPV.0000000000001127. Epub 2022 Jan 12. PMID 35030139
- [Background] Mari JJ, Williams P. A comparison of the validity of two psychiatric screening questionnaires (GHQ-12 and SRQ-20) in Brazil, using Relative Operating Characteristic (ROC) analysis. Psychol Med. 1985 Aug;15(3):651-9. doi: 10.1017/s0033291700031500. PMID 4048323
- [Background] Krhut J, Gartner M, Mokris J, Horcicka L, Svabik K, Zachoval R, Martan A, Zvara P. Effect of severity of urinary incontinence on quality of life in women. Neurourol Urodyn. 2018 Aug;37(6):1925-1930. doi: 10.1002/nau.23568. Epub 2018 Mar 31. PMID 29603780
- [Background] D'Ancona C, Haylen B, Oelke M, Abranches-Monteiro L, Arnold E, Goldman H, Hamid R, Homma Y, Marcelissen T, Rademakers K, Schizas A, Singla A, Soto I, Tse V, de Wachter S, Herschorn S; Standardisation Steering Committee ICS and the ICS Working Group on Terminology for Male Lower Urinary Tract & Pelvic Floor Symptoms and Dysfunction. The International Continence Society (ICS) report on the terminology for adult male lower urinary tract and pelvic floor symptoms and dysfunction. Neurourol Urodyn. 2019 Feb;38(2):433-477. doi: 10.1002/nau.23897. Epub 2019 Jan 25. PMID 30681183
- [Background] Wexner SD, Bleier J. Current surgical strategies to treat fecal incontinence. Expert Rev Gastroenterol Hepatol. 2015;9(12):1577-89. doi: 10.1586/17474124.2015.1093417. Epub 2015 Sep 28. PMID 26414494
- [Background] Bharucha AE, Dunivan G, Goode PS, Lukacz ES, Markland AD, Matthews CA, Mott L, Rogers RG, Zinsmeister AR, Whitehead WE, Rao SS, Hamilton FA. Epidemiology, pathophysiology, and classification of fecal incontinence: state of the science summary for the National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) workshop. Am J Gastroenterol. 2015 Jan;110(1):127-36. doi: 10.1038/ajg.2014.396. Epub 2014 Dec 23. PMID 25533002
- [Background] Menees S, Chey WD. Fecal Incontinence: Pathogenesis, Diagnosis, and Updated Treatment Strategies. Gastroenterol Clin North Am. 2022 Mar;51(1):71-91. doi: 10.1016/j.gtc.2021.10.005. Epub 2022 Jan 7. PMID 35135666